CLINICAL TRIAL: NCT04613505
Title: Determining Parental Attitudes Toward Day of Surgery Consent for Research
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Katherine Taylor, Staff Anesthesiologist, The Hospital for Sick Children
Other Study IDs: 1000066221
Record Dates: First submitted 2020-10-02; First posted 2020-11-03 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Surgery; Consent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Phase 1: Instrument Development: Parents will be asked to participate in a semi-structured interview with one of the researchers that will explore their attitudes toward day of surgery consent. Particular attention will be given to a) study designs, b) previous research experience, and c) previous medical experiences.
  Interventions: Behavioral: Semi-structured interview
- Phase 2: Questionnaire Adaptation: Parents will be given approximately 5 minutes to review a questionnaire we developed using participant responses in Phase 1. After reviewing the questionnaire, participants will be asked to participate in a semi-structured interview with one of the investigators.
  Interventions: Behavioral: Semi-structured interview
- Phase 3: Questionnaire Application & Development of Day of surgery consent Table of Guidelines: Participants will be asked to complete the questionnaire developed in Phase 2.
  Interventions: Behavioral: Same day consent questionnaire
- Phase 4: Table of Guidelines Refinement: Participants will be given approximately 5 minutes to review the table of guidelines developed in Phase 3. After reviewing the guidelines, participants will be asked to participate in a semi-structured interview with one of the investigators.
  Interventions: Behavioral: Semi-structured interview

INTERVENTIONS:
Behavioral: Semi-structured interview — Participants will be asked a set of questions as applicable to each phase. Researchers will be able to ask additional questions as they arise within each interview.
  Groups: Phase 1: Instrument Development; Phase 2: Questionnaire Adaptation; Phase 4: Table of Guidelines Refinement
Behavioral: Same day consent questionnaire — A questionnaire (yet to be developed) will be administered to participants.
  Groups: Phase 3: Questionnaire Application & Development of Day of surgery consent Table of Guidelines

SUMMARY:
There are no studies examining parents' attitudes towards day of surgery consent for research. The purpose of the study is to determine the attitudes parents of potential research participants have toward being approached for day of surgery consent. The primary objective is to determine parental attitudes regarding day of surgery consent for anesthesia research. The secondary objective is to determine the boundaries for day of surgery consent (e.g., study types, interventions, risk factors).

DETAILED DESCRIPTION:
This is a multi-phase prospective cohort study. In the first phase the investigators will interview parents and consult the Family Research Advisory Committee (FRAC) to determine their attitudes toward day of surgery research consent. The investigators will use the participants' responses and instruments already found in the literature to develop the questionnaire. In the second phase, the investigators will interview parents and consult FRAC about the questionnaire to determine which items to add, remove, or modify. In the third phase, the investigators will distribute the adapted questionnaire to clarify parents' attitudes surrounding day of surgery consent. The investigators will use the results of the third phase to develop a table of guidelines for day of surgery consent. In the final phase, the investigators will interview parents, healthcare professionals, and consult FRAC for feedback and modification of the table of guidelines.

ELIGIBILITY:
Inclusion Criteria:

* The parents of children undergoing elective surgical procedures at Sickkids will be invited to participate in the study.
* If multiple parents are present, they are permitted to participate jointly; however, their participation will count as a single response.

Exclusion Criteria:

-Parents of children who are undergoing urgent or add-on procedures will be excluded.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All participants receiving same day surgery at our institution are eligible to participate.
Sampling Method: Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Parental attitude towards day of surgery consent | Day of surgery
  Semi-structured interviews

SECONDARY OUTCOMES:
Boundary for day of surgery consent | Day of surgery
  Semi-structured interview
Boundary for day of surgery consent | Day of surgery
  Questionnaires to be developed in phases 1 and 2 of the study

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Taylor, Principal Investigator — Staff Anesthesiologist
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No